CLINICAL TRIAL: NCT02989129
Title: Prospective Open Labeled Pilot Trial of Quercetin in the Treatment and Prevention of Chemotherapy-induced Neuropathic Pain in Cancer Patients
Brief Title: Trial of Quercetin in the Treatment and Prevention of Chemotherapy-induced Neuropathic Pain in Cancer Patients
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: FDA IND Approval
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0287
Record Dates: First submitted 2016-12-08; First posted 2016-12-12 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Polyneuropathies and Other Disorders of the Peripheral Nervous System; Chemotherapy Induced Neuropathic Pain
Keywords: Polyneuropathies and Other Disorders of the Peripheral Nervous System; Chemotherapy Induced Neuropathic Pain; CINP; Quercetin; Questionnaires; Surveys
MeSH Terms: conditions — Polyneuropathies | interventions — Surveys and Questionnaires; Quercetin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Chemotherapy Induced Neuropathic Pain (CINP) Treatment Group (Experimental): Questionnaires completed at Baseline and at End of Study Visit.
  Participants take Quercetin tablets by mouth 2 times every day for 12 weeks.
  Interventions: Behavioral: Questionnaires; Drug: Quercetin
- Chemotherapy Induced Neuropathic Pain (CINP) Prevention Group (Experimental): Questionnaires completed at Baseline and at End of Study Visit.
  Participants take Quercetin tablets by mouth 2 times every day for 12 weeks.
  Interventions: Behavioral: Questionnaires; Drug: Quercetin

INTERVENTIONS:
Behavioral: Questionnaires — Questionnaires regarding quality of life, pain level, and related symptoms completed at Baseline and at End of Study Visit.. It should take less than 1 hour to complete these questionnaires.
  Other Names: Surveys
Drug: Quercetin — 500 mg by mouth twice daily (after breakfast and dinner) for 12 weeks during study.

SUMMARY:
The goal of this clinical research study is to learn about the effectiveness of quercetin in treating and preventing CINP. Researchers also want to learn if quercetin has an effect on participant's quality of life.

DETAILED DESCRIPTION:
Study Product Administration:

If participant is found to be eligible to take part in this study, participant will take quercetin tablets by mouth 2 times every day for 12 weeks. The study staff will give participant the tablets and additional instructions on how to take the study product.

Length of Participation:

Participant may take quercetin for up to 12 weeks. Participant will no longer be able to take quercetin if the pain symptoms gets worse, if intolerable side effects occur, or if participant is unable to follow study directions.

Study Visits:

Every week, participant will either come to the clinic or a member of the staff will call participant to learn how participant is doing, if participant has had any side effects, and to check that participant is taking quercetin correctly. Participant will also complete a questionnaire about any pain symptoms participant may be having. The call/questionnaire should take about 10-15 minutes to complete.

End-of-Study Visit:

About 7 days after participant's last dose of quercetin, participant will complete the same questionnaires participant completed at screening.

Participation in this study will be over after the end-of-study visit.

This is an investigational study. Quercetin is commercially available as a supplement, but it is not FDA approved.The study doctor can explain how the study product is designed to work.

Up to 20 participants will be enrolled in this study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients > 18 years old.
2. Patients starting, undergoing or completed chemotherapy at MD Anderson Cancer Center
3. Any cancer patients who received any of the chemotherapeutic agents listed below and developed neuropathic pain for the treatment cohort; or any cancer patients who have been scheduled to receive any of the chemotherapeutic agents listed below for the preventive cohort. The chemotherapeutic agents include 1) taxanes (paclitaxel, docetaxel), 2) vinca alkaloids (vincristine, vinblastine), 3) platinum agents (cisplatin, carboplatin, oxaliplatin), and 4) others (thalidomide, bortezomib, lenalidomide).
4. Patients have neuropathic pain intensity of at least 4/10 on numeric rating score (NRS, 0/10 being no pain and 10/10 excruciating pain) for the treatment cohort; or 0/10 on NRS for the preventive cohort.
5. Patients are on stable dose of any medication
6. Patients followed at the Pain Medicine department. Patients with normal renal function (Normal values, BUN (blood urea nitrogen): 8 to 20 mg/dL, Creatinine: 0.7 to 1.3 mg/dL).
7. Patients able to speak English.
8. Patients able to review, understand, and provide written consent.
9. Patients with an Eastern Cooperative Oncology performance (ECOG) status of 0-2.

Exclusion Criteria:

1. Renal impairment.
2. Pregnancy.
3. Hypersensitivity reaction, anaphylaxis, or any other serious adverse reaction to quercetin or product components.
4. Patients who are enrolled in another Pain Medicine trial.
5. Patients with malabsorption syndrome or resection of the stomach or small bowel.
6. Patients with any condition that precludes use of the study medication as determined by the treating physician.
7. Patients taking Quercetin for other medical reasons.
8. Patients taking Digoxin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-04 (Estimated); Primary Completion 2020-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Change in Neuropathic Pain Intensity | 12 weeks
  Primary endpoint is the change in neuropathic pain intensity during 12 weeks of treatment using the the Douleur Neuropathique en 4 questions (DN4).

CONTACTS AND LOCATIONS:
Overall Officials: Salahadin Abdi, MD, PHD, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org